CLINICAL TRIAL: NCT00867906
Title: A Double-blind, Randomised, Placebo-controlled Study to Assess the Safety of Cat-PAD in Cat Allergic Subjects With Controlled Asthma
Brief Title: Safety of Cat-PAD to Treat Cat Allergy in Cat Allergic Subjects With Controlled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Dr Rod Hafner, Circassia Limited
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP003
Record Dates: First submitted 2009-03-19; First posted 2009-03-24 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Cat Allergy
Keywords: Cat allergy; Immunotherapy; Cat-PAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Other): Asthmatics using salbutamol only, subjects to receive either Cat-PAD or placebo comparator
  Interventions: Biological: Cat-PAD; Biological: Placebo
- Cohort 2 (Other): Asthmatics using inhaled corticosteroid, subjects to receive either Cat-PAD or placebo comparator
  Interventions: Biological: Cat-PAD; Biological: Placebo
- Cohort 3 (Other): Asthmatics using inhaled corticosteroid and LABA, subjects to receive either Cat-PAD or placebo comparator
  Interventions: Biological: Cat-PAD; Biological: Placebo

INTERVENTIONS:
Biological: Cat-PAD — Cat-PAD dose 1x8 administrations 2 weeks apart
Biological: Placebo — Placebo comparator, 1x8 administrations 2 weeks apart

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis and/or asthma. Cat-PAD is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of cat allergy.

This study will evaluate the safety and tolerability of multiple doses of Cat-PAD in controlled asthmatics treated with either inhaled salbutamol, inhaled corticosteroids or inhaled corticosteroids with a LABA and to explore the efficacy of Cat-PAD in these subjects using the Late Phase Skin Response, Early Phase Skin Response, and Conjunctival Provocation Test.

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled, parallel group, multiple dose study to evaluate the safety and tolerability of Cat-PAD in cat allergic subjects with allergic rhinoconjunctivitis and controlled asthma. The efficacy of Cat-PAD will also be explored in these subjects using the EPSR, LPSR, CPT, and levels of cat specific IgE. A single centre will be initiated first, with a second centre included as a backup, if needed, to enable recruitment numbers to be met.

Three cohorts will be studied, depending on the treatment used to control the subject's asthma:Cohort 1 - inhaled salbutamol only, Cohort 2 - inhaled corticosteroid only, Cohort 3 - inhaled corticosteroid plus a LABA

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 8 weeks before randomisation and may consist of one or two visits to the clinic, at the investigator's discretion. Baseline Challenge will consist of a single visit 1 to 4 weeks before randomisation.

In Period 2, subjects in each cohort complying with the inclusion/exclusion criteria will be randomised to either 3 nmol Cat-PAD or placebo. Treatments will be administered every 2 weeks (±2 days) for 14 week

In Period 3, Post Treatment Challenge consist of a single visit 24-28 weeks after the first administration in the treatment period and assessments will be performed identical to those at the baseline challenge. Follow-up will be conducted 3-10 days after PTC.

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged 18-65 years.
* A history of controlled asthma as defined in GINA (2007) on exposure to cats for at least 1 year
* Asthma controlled with:Inhaled salbutamol (Cohort 1), Inhaled corticosteroid (Cohort 2), Inhaled corticosteroid plus a long acting β2agonist (LABA) (Cohort 3) Treatment for asthma must have been stable (drug(s), dose, frequency) for at least 3 months.
* A reliable history of rhinoconjunctivitis (sneezing, rhinorrhoea, nasal blockage, itchy/red/sore/watering eyes) on exposure to cats for at least 1 year.
* Subjects who provide written informed consent.
* Positive skin prick test to cat allergen with a wheal diameter at least 3mm larger than that produced by the negative control.
* A LPSR to cat allergen eight hours after intradermal injection of greater than 25mm diameter.
* Positive CPT with a score ≥4.
* The subject must be willing and able to comply with the study requirements.
* If the subject is female and of childbearing potential she must practice an acceptable form of contraception, and produce a negative urine pregnancy test on the Screening Visit. A female subject may be included without a negative urine pregnancy test if she can document that she is surgically sterile or at least 2 years post-menopausal.

Exclusion Criteria

* Subjects with asthma falling under GINA (2007) definitions "partly controlled" and "uncontrolled"
* Subjects with a requirement for more than 1000 µg beclomethasone (or equivalent) per day for the treatment of asthma.
* A history of anaphylaxis to cat allergen.
* Subjects with a cat specific IgE >100 kU/L.
* Subjects with an FEV1 <80% of normal
* Subjects with an acute phase skin response to cat allergen with a wheal diameter > 30mm.
* Subjects who suffer from seasonal allergic rhinoconjunctivitis, and cannot complete the baseline/post-treatment challenge (PTC) and the dosing periods outside the respective pollen season.
* Allergen immunotherapy during the last 12 months or any history of Cat Dander immunotherapy.
* Subjects who have completed or are undergoing ongoing treatment with anti-IgE-antibody.
* Use of the therapies listed in Section 5.9.2 at any time during the study will make the subject ineligible for the study.
* The subject has unacceptable symptoms in the 3 days without loratadine prior to the screening visit.
* Subjects for whom administration of adrenaline is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* Subjects being treated with beta-blockers.
* Have symptoms of a clinically relevant illness in the Investigator's opinion, within 6 weeks prior to Screening Visit.
* Female subjects who are pregnant, lactating or planning a pregnancy during the study.
* Have any clinically relevant abnormalities detected on physical examination.
* 12-lead ECG or vital signs (blood pressure, pulse rate, respiratory rate and oral temperature) that are outside normal limits, unless the abnormality is considered not to be of clinical relevance by the Investigator.
* Laboratory values (haematology, biochemistry, urine tests) that are outside the normal ranges, unless the abnormality is considered not to be of clinical relevance by the Investigator.
* Significant history of alcohol or drug abuse.
* History of immunopathological diseases.
* Positive test for hepatitis B, hepatitis C or HIV at screening.
* Previously randomised into this study or have received Cat-PAD (or a prototype thereof) previously.
* Have a history of severe drug allergy or anaphylactic reaction to food.
* Planned travel outside the study area for a substantial portion of the study period.
* Have received treatment with an investigational drug within 6 months prior to study screening or have participated in a study with a new formulation of a marketed drug one month prior to study screening.
* Are unable to communicate or to understand the requirements of the study, or any psychiatric disorder, which would impair communication between the subject and the Investigator thereby interfering with the informed consent procedure or the gathering of study data.
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study.
* Subjects with a known allergy to thioglycerol.
* Subjects who have a dependent relationship (e.g. employees or family members) with either the Sponsor or Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple intradermal injections of Cat-PAD in cat allergic subjects with controlled asthma | 28 weeks

SECONDARY OUTCOMES:
Mean change from baseline in area of the LPSR 8 hours after intradermal challenge with whole cat allergen at PTC after Cat-PAD injection compared to placebo | 28 weeks
Mean change from baseline in area of the EPSR 15 minutes after intradermal challenge with whole cat allergen at PTC after Cat-PAD injection compared to placebo | 28 weeks
Mean change from baseline in CPT score at PTC after Cat-PAD injection compared to placebo | 28 weeks
Mean change from baseline in concentration of cat specific IgE at PTC after Cat-PAD injection compared to placebo | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amarjit Cheema, MD, Principal Investigator — Alpha Medical Research
Locations (1):
- Alpha Medical Research, Mississauga, Toronto, Ontario, Canada